CLINICAL TRIAL: NCT04885920
Title: Prospective, Non-interventional, Observational Study in Patients With IBD Receiving IV or SC Vedolizumab Therapy to Observe Route of Administration Choices and Outcomes
Brief Title: A Study on Administration Choices of Vedolizumab and Outcomes for Adults With Inflammatory Bowel Disease (IBD) (VARIETY - CROATIA AND SLOVENIA)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4036
Record Dates: First submitted 2021-05-12; First posted 2021-05-13 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Crohns Disease; Colitis, Ulcerative
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With IBD: Participants diagnosed with moderately to severely active IBD (UC or CD) who initiated or are currently ongoing vedolizumab IV induction treatment in accordance with the current Summary of Product Characteristics (SmPC) or receiving vedolizumab ongoing or maintenance IV treatment with the option to switch to vedolizumab SC treatment, will be observed prospectively for at least 12 months.

SUMMARY:
Inflammatory bowel disease consists of either ulcerative colitis (UC) or Crohn's disease (CD).

The main aim of this study is to describe real-world treatment patterns in adults with moderate to severe ulcerative colitis or Crohn's disease when treated with vedolizumab. This will include the administration choices which can either be an infusion through a vein (intravenous or IV), or an injection just under the skin (subcutaneous injection, or SC).

Treatment will be determined by the study doctor according to routine clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with IBD who initiated or who are currently ongoing induction or maintenance with vedolizumab in the real world setting.

The study will enroll approximately 120 participants. The data will be collected prospectively at the study sites and will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

* Participants with IBD

This multi-center study will be conducted in Croatia and Slovenia having specialized gastroenterology centers. The overall duration of the study will be at least 26 months. Data will be collected at baseline, at 3 months (+/- 1 month) after induction, and every 6 months (+/- 1 month) after that, and at the time of switch, discontinuation and/or at routine follow-up visits up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has moderately to severely active IBD (UC or CD), initiating or ongoing IV induction treatment with vedolizumab in accordance with the current SmPC at baseline OR IBD participants receiving ongoing/maintenance IV vedolizumab treatment, with the option to switch to SC vedolizumab maintenance treatment.

Exclusion Criteria:

1. Prior history of intolerability, hypersensitivity, or other contraindications (active severe infections such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as Progressive Multifocal Leukoencephalopathy) to vedolizumab therapy as defined in the current SmPC.
2. Current or planned participation in an interventional clinical trial for CD or UC.
3. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active UC or CD receiving vedolizumab treatment in accordance with the approved SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Persisting to Treatment With Vedolizumab IV Compared to Participants With Treatment Change at 12 Months | Baseline up to 12 months
Time to any Treatment Change | Baseline up to 12 months
Number of Participants With Reason for Treatment Change | Baseline up to 12 months
Number of Participants With Change in Vedolizumab Dosing Frequency | Baseline up to 12 months
Number of Participants Who Discontinued the Vedolizumab Treatment | Baseline up to 12 months
Number of Participants Who Changed to Another Treatment | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Croatia (5):
  - Klinicki bolnicki centar Osijek (University medical centre Osijek), Osijek
  - Klinicki bolnicki centar Rijeka (University medical centre Rijeka), Rijeka
  - Klinicki bolnicki centar Split (University medical centre Split), Split
  - Klinicki bolnicki centar Sestre milosrdnice (University medical centre Sestre milosrdnice), Zagreb
  - Klinicki bolnicki centar Zagreb (University medical centre Zagreb), Zagreb
- Slovenia (3):
  - Splosna bolnisnica Celje (General hospital Celje), Celje
  - Univerzitetni klinicni center Ljubljana (University medical Centre Ljubljana), Ljubljana
  - Univerzitetni klinicni center Maribor (University medical centre Maribor), Maribor

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60a2b6c1ef0b71001e743cb7